CLINICAL TRIAL: NCT04352062
Title: The Usefulness of Melatonin Supplementation in Postmenopausal Women With Helicobacter Pylori-associated Dyspepsia
Brief Title: Melatonin Supplementation in Postmenopausal Women With H. Pylori-associated Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMWH-D-20-00081
Record Dates: First submitted 2020-03-09; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-03

CONDITIONS: Melatonin Deficiency
MeSH Terms: interventions — Melatonin; Pantoprazole; Amoxicillin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Group (Experimental): Melatonin ( 5-Methoxy-N-Acetyltryptamine) at dose 1mg/morning and 3mg/at bedtime (period 6 months)
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): 1 tablet twice daily (period 6 months)
  Interventions: Other: placebo
- Helicobacter pylori infected group (Other): Pantoprazole 2 x 40mg (twice daily) Amoxicyllin 2 x 1000mg (twice daily) Lovofloxacin 2 x 500mg (twice daily)
  Interventions: Drug: Pantoprazole 40mg; Drug: Amoxicillin; Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Melatonin
  Arms: Treatment Group
Other: placebo
  Arms: Placebo
Drug: Pantoprazole 40mg — pantoprazole 2 x 40mg
  Other Names: Pantoprazole
  Arms: Helicobacter pylori infected group
Drug: Amoxicillin — Amoxicillin 2 x 1000mg
  Other Names: Amoxycillin
  Arms: Helicobacter pylori infected group
Drug: Levofloxacin 500mg — Levofloxacin 2 x 500mg
  Other Names: Levofloxacin
  Arms: Helicobacter pylori infected group

SUMMARY:
Background: The aim of the study was to assess the role of melatonin in chronic dyspepsia in this group of women, with consideration of Helicobacter infection. Methods: The study comprised 152 subjects Including 30 healthy women (group I), 60 women with asymptomatic H.pylori infection (group II), and 64 women H. pylori infected with chronic dyspepsia(group III). Endoscopic examination, histological assessment of gastric end duodenal mucosa, urease breath test(UBT-13C), and serum levels of 17-β-estradiol, follicle stimulating hormone, melatonin and urinary concentration of 6-sulfatoxymelatonin were determined by immunoenzymatic method. In group III - 14-day antibacterial treatment was introduced with pantoprazole, amoxicillin and levofloxacin. Afterward, in 32 women was administered placebo(group IIIa), and in 32 women (group IIIb) melatonin at a dose 1 m/morning and 3 mg/at bedtime, for six months.

DETAILED DESCRIPTION:
Background:Dyspeptic syndrome in the form of epigastric pain are particularly frequent in postmenopausal women. The aim of the study was to assess the role of melatonin in chronic dyspepsia in this group of women, with consideration of Helicobacter infection. Methods: The study comprised 152 subjects Including 30 healthy women (group I), 60 women with asymptomatic H.pylori infection (group II), and 64 women H. pylori infected with chronic dyspepsia(group III). Endoscopic examination, histological assessment of gastric end duodenal mucosa, urease breath test(UBT-13C), and serum levels of 17-β-estradiol, follicle stimulating hormone, melatonin and urinary concentration of 6-sulfatoxymelatonin were determined by immunoenzymatic method. In group III - 14-day antibacterial treatment was introduced with pantoprazole, amoxicillin and levofloxacin. Afterward, in 32 women was administered placebo(group IIIa), and in 32 women (group IIIb) melatonin at a dose 1 m/morning and 3 mg/at bedtime, for six months.

ELIGIBILITY:
Inclusion Criteria:

Patients with

* Epigastric pain of a hunger nature
* Pain at night in the epigastric region
* Increased appetite

Exclusion Criteria:

Patients with

* Functional or inflammatory diseases of the gastrointestinal tract liver and pancreas
* Metabolic, allergic and mental disease
* Hormone replacement therapy

Ages: 49 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2011-01-09 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
10 point Visual Analogue Scale (VAS) of Dyspeptic symptoms | 6 months
  scale that access severity of Dyspeptic symptoms such as: epigastric pain of hunger nature and pain in the epigastric region at night (intensity measured from 1 to 10 points)

CONTACTS AND LOCATIONS:
Overall Officials: Cezary Chojnacki, MD.PhD., Principal Investigator — Department of Clinical Nutrition and Gastroenterological Diagnostics
Locations (1):
- Department of Clinical Nutrition and Gastroenterological Diagnostics Medical University of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heinemann LA, Potthoff P, Schneider HP. International versions of the Menopause Rating Scale (MRS). Health Qual Life Outcomes. 2003 Jul 30;1:28. doi: 10.1186/1477-7525-1-28. PMID 12914663
- [Derived] Chojnacki C, Medrek-Socha M, Konrad P, Chojnacki J, Blonska A. The value of melatonin supplementation in postmenopausal women with Helicobacter pylori-associated dyspepsia. BMC Womens Health. 2020 Nov 26;20(1):262. doi: 10.1186/s12905-020-01117-z. PMID 33243209